CLINICAL TRIAL: NCT02051985
Title: Early-start Exercise Training After Acute Hemodynamic Decompensation in Patients With Chronic Heart Failure. A Multicenter, Randomized, Controlled Trial on Feasibility and Impact on Functional Capacity, Symptoms and Neurohumoral Activation.
Brief Title: Early-start Exercise Training in Subacute Heart Failure
Acronym: RE-START
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione Salvatore Maugeri (Other)
Responsible Party: Principal Investigator, Alessandro Mezzani, MD, Fondazione Salvatore Maugeri
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEC 877
Record Dates: First submitted 2014-01-29; First posted 2014-01-31 (Estimated); Last update posted 2014-01-31 (Estimated); Status verified 2014-01

CONDITIONS: Chronic Heart Failure; Heart Decompensation
Keywords: Chronic heart failure; Heart decompensation; Aerobic exercise training; Functional capacity; Dyspnea; Beta-adrenergic receptor signaling
MeSH Terms: conditions — Heart Failure; Dyspnea

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aerobic exercise training (Experimental)
  Interventions: Other: Aerobic exercise training
- Standard physical therapy (Active Comparator)
  Interventions: Other: Standard physical therapy

INTERVENTIONS:
Other: Aerobic exercise training — Days 1-2: active assisted mobilization (2 sessions/day, each 30 minutes duration).
  Days 3-4: as days 1-2 + unloaded bedside cycle ergometer (3 sessions/day, each 5-6 minutes duration).
  Days 5-6: as days 1-2 + bedside cycle ergometer at 10 W (3 sessions/day, each 15-20 minutes duration).
  Days 7-12: as days 1-2 + bedside cycle ergometer at 10-20 W (3 sessions/day, each 15-20 minutes duration).
  In addition, when possible according to their clinical conditions, patients will undergo one assisted ambulation session of 15-20 minutes per day.
  Arms: Aerobic exercise training
Other: Standard physical therapy — Days 1-2: active assisted mobilization (2 sessions/day, each 30 minutes duration).
  Days 3-12: active assisted mobilization (1 session/day, 30 minutes duration).
  In addition, when possible according to their clinical conditions, patients will undergo one assisted ambulation session of 15-20 minutes per day.
  Arms: Standard physical therapy

SUMMARY:
The purpose of this study is to evaluate the feasibility and the short-term effects of an early-start aerobic exercise training program on functional capacity, symptoms and neurohormonal activation in chronic heart failure patients with recent acute hemodynamic decompensation.

DETAILED DESCRIPTION:
Prescription of aerobic exercise training in stable chronic heart failure patients finds an evidence-based justification in the acknowledged long-term positive effects of aerobic exercise training on both functional capacity and prognosis in this population. In recent time, evidence has accumulated in normal subjects about short-term favorable effects of aerobic exercise training on sympatho-vagal balance and flow-mediated vasodilation, two physiological mechanisms known to be profoundly altered in the setting of acute hemodynamic decompensation of chronic heart failure. The possible extension of aerobic exercise training indication to chronic heart failure patients admitted for recent acute hemodynamic decompensation not stabilized as yet, may thus provide a valuable, low-cost tool to effectively manage such a high-risk and resource-absorbing population.

ELIGIBILITY:
Inclusion Criteria:

* history of chronic heart failure for at least 6 months, with ongoing acute decompensation defined as onset or worsening of heart failure signs and/or symptoms during the previous 15 days with need of intravenous diuretic and/or vasodilator therapy;
* age >18 years
* left ventricular ejection fraction <40%
* proBNP >1000 pg/ml at admission

Exclusion Criteria:

* ongoing cardiogenic shock
* need of intravenous inotropic therapy
* acute coronary syndrome during the preceding 3 months
* clinical and/or instrumental evidence of myocardial ischemia and/or life-threatening arrhythmias
* previous cardiac valve surgery
* creatinine >2.5 mg/dl at admission
* severe comorbidities limiting functional capacity

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2013-10; Primary Completion 2015-06 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Distance walked at 6-min walking test | 12 days of intervention
  Change from baseline in distance walked at 6-min walking test

SECONDARY OUTCOMES:
Aerobic exercise training safety and tolerability | 12 days of treatment
  Number of participants with serious/non-serious adverse events and completing/not completing the study protocol
Patient-reported dyspnea, evaluated by a 7-point Likert scale | 12 days of intervention
  Change from baseline in patient-reported dyspnea on a 7-point Likert scale
Levels of lymphocyte G protein-coupled receptor kinase-2 | 12 days of intervention
  Change from baseline in lymphocyte G protein-coupled receptor kinase-2 levels
Levels of circulating inflammatory and angiogenetic markers (TNF-alfa, Interleukin-6, Angiopoietin 2 and VEGF) | 12 days of intervention
  Change from baseline in circulating inflammatory and angiogenetic markers (TNF-alfa, Interleukin-6, Angiopoietin 2 and VEGF) levels

CONTACTS AND LOCATIONS:
Overall Officials: Pantaleo Giannuzzi, MD, Study Chair — Fondazione Salvatore Maugeri - Scientific Institute of Veruno; Alessandro Mezzani, MD, Principal Investigator — Fondazione Salvatore Maugeri - Scientific Institute of Veruno
Locations (9):
- Italy (9):
  - Fondazione Salvatore Maugeri, IRCCS - Scientific Institute of Cassano Murge, Cassano Murge
  - Fondazione Salvatore Maugeri, IRCCS - Scientific Institute of Lumezzane, Lumezzane
  - Fondazione Salvatore Maugeri - Scientific Institute of Milano, Milan
  - Fondazione Salvatore Maugeri, IRCCS - Scientific Institute of Montescano, Montescano
  - Fondazione Salvatore Maugeri, IRCCS - Scientific Institute of Pavia, Pavia
  - Fondazione Salvatore Maugeri, IRCCS - Scientific Institute of Telese Terme, Telese Terme
  - Fondazione Salvatore Maugeri - Presidio Major of Torino, Torino
  - Fondazione Salvatore Maugeri, IRCCS - Scientific Institute of Tradate, Tradate
  - Fondazione Salvatore Maugeri, IRCCS - Scientific Institute of Veruno, Veruno

REFERENCES:
- See also: Related Info — http://www.fsm.it